CLINICAL TRIAL: NCT06044675
Title: A Randomized Trial of MDMA-Assisted Cognitive-Behavioural Conjoint Therapy (CBCT) Versus CBCT in Dyads in Which One Member Has Posttraumatic Stress Disorder (PTSD)
Brief Title: MDMA-Assisted CBCT for PTSD vs CBCT RCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Remedy (Industry)
Collaborators: Remedy Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ICAPT1
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Post Traumatic Stress Disorder
Keywords: MDMA; Cognitive Behavioural Conjoint Therapy (CBCT); Relationship functioning
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MDMA-Assisted CBCT Condition (Experimental): Dyads will undergo a 7-week course of CBCT psychotherapy for PTSD with two sessions that integrate MDMA-assisted psychotherapy. MDMA will be administered in two separate sessions and integrated into the psychotherapy protocol. The two doses of MDMA during this study will be used as an adjunct to psychotherapy.
  Interventions: Drug: MDMA assisted psychotherapy
- CBCT-Only Condition (Active Comparator): Dyads will undergo a 7-week course of CBCT psychotherapy for PTSD. Dyads who have undergone the CBCT-Only condition will have the option to do a crossover and have the two MDMA sessions after follow-up.
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Drug: MDMA assisted psychotherapy — This treatment combines MDMA with a well researched treatment for PTSD for dyads known as CBCT. Dyads will undergo a 7-week course of psychotherapy with two doses of MDMA will be used as an adjunct to psychotherapy.
  Other Names: MDMA-assisted CBCT
  Arms: MDMA-Assisted CBCT Condition
Behavioral: Psychotherapy — A manualized treatment for PTSD for dyads wherein one person has symptoms of PTSD. This intervention is 7-week course of psychotherapy that is designed to simultaneously improve PTSD symptoms and relationship functioning through education and skill training.
  Other Names: CBCT
  Arms: CBCT-Only Condition

SUMMARY:
This study aims to evaluate the safety, feasibility, acceptability, and effectiveness of MDMA-assisted Cognitive-Behavioral Conjoint Therapy (CBCT) versus CBCT alone for the treatment of Post-Traumatic Stress Disorder (PTSD). PTSD is a debilitating condition that significantly impacts interpersonal relationships and the functioning of individuals and their loved ones. There is also a well-established reciprocal relationship between interpersonal relationships, PTSD, and recovery.

CBCT is a manualized treatment for PTSD that simultaneously addresses PTSD symptoms and relationship satisfaction. It provides dyads with behavioral tools to navigate PTSD-related challenges, as well as the knowledge behind PTSD and how it impacts relationships. Previous research has demonstrated the efficacy of CBCT in improving PTSD symptoms, partner functioning, and relationship satisfaction in both distressed and non-distressed dyads.

MDMA is a drug commonly used recreationally that has been increasingly studied because of its ability to reduce the impact of PTSD symptoms. The effects of MDMA are reduced fear, enhanced communication, trust and introspection, and increased empathy and compassion. The effects of MDMA create a state that enhances the positive effects of therapy by increasing the ability to tolerate negative emotions and allowing clients to stay engaged in therapy without being overwhelmed by the intense emotions surrounding the memories of traumatic events. It is believed that MDMA may help promote the effects of CBCT due to its ability to induce empathy and interpersonal openness.

This randomized study is the second study designed to explore the efficacy of combining MDMA-assisted therapy with CBCT. This study will enroll 30 dyads, where one individual has symptoms of PTSD. Participants will undergo a 7-week psychotherapy course, in MDMA-assisted CBCT or CBCT alone. In the MDMA-assisted CBCT, participants will go through CBCT sessions, and two doses of MDMA will be used as an adjunct to psychotherapy. Participants assigned to the CBCT-only condition will go through CBCT sessions and will have the opportunity to crossover and receive the two MDMA sessions after follow-up. The primary goal of this research is to contribute to the literature on MDMA-assisted CBCT by investigating its feasibility, safety, acceptability, and effectiveness, and by comparing it to active PTSD treatments.

ELIGIBILITY:
Inclusion Criteria

* Participant with PTSD

  1. Participant with PTSD
  2. Meet criteria for PTSD
  3. Have a close other person who is able and willing to participate in this study
  4. Are at least 18 years old
  5. Are a resident of Ontario and live within the Greater Toronto Area (GTA)
  6. Are in good physical health
  7. Are proficient in speaking and reading English
  8. Are willing to have all visits audio and video recorded
  9. Are able to swallow pills
  10. Agree to all study rules and commit to all medical and therapy visits
  11. If in psychotherapy, are willing to allow the study therapists to communicate directly with your therapist
  12. Are willing to stop taking psychiatric medications, herbal supplements, prescription and nonprescription medications during the study
  13. Agree to stay overnight on two separate occasions after each full-day MDMA-Assisted Therapy Session, and not to drive for at least 24 hours after taking MDMA
  14. Are not pregnant and will commit to not becoming pregnant during the study, if you are able to become pregnant
  15. Have a supportive relative, spouse, close friend or other caregiver not participating in this study who can serve as your emergency contact
  16. Agree to inform the researchers within 48 hours of any medical conditions and procedures
  17. Agree to not participate in any other clinical trials during this study
* Close Significant Other

  1. Have a close other person who meets criteria for PTSD and is able and willing to participate in this study
  2. Are at least 18 years old
  3. Are a resident of Ontario and live within the Greater Toronto Area (GTA)
  4. Are in good physical health
  5. Are proficient in speaking and reading English
  6. Are willing to have all visits audio and video recorded
  7. Are able to swallow pills
  8. Agree to all study rules and commit to all medical and therapy visits
  9. If in psychotherapy, are willing to allow the study therapists to communicate directly with your therapist
  10. Are willing to stop taking psychiatric medications, herbal supplements, prescription and nonprescription medications during the study
  11. Agree to stay overnight on two separate occasions after each full-day MDMA-Assisted Therapy Session, and not to drive for at least 24 hours after taking MDMA
  12. Are not pregnant and will commit to not becoming pregnant during the study, if you are able to become pregnant
  13. Have a supportive relative, spouse, close friend or other caregiver not participating in this study who can serve as your emergency contact
  14. Agree to inform the researchers within 48 hours of any medical conditions and procedure
  15. Agree to not participate in any other clinical trials during this study

Exclusion Criteria

* Participant with PTSD

  1. Are pregnant or could become pregnant and not using birth control
  2. Have a history of, or a current psychotic disorder or bipolar 1 disorder or dissociative identity disorder
  3. Have a history of a medical condition that could make receiving MDMA unsafe (e.g. glaucoma, heart attack, stroke, aneurysm)
  4. Have a history of Diabetes Mellitus (Type 2) that a doctor determines is not stable
  5. Have hypothyroidism (low activity in the thyroid gland) and are not on thyroid replacement
  6. Have high blood pressure, a history of heart disease, heart failure, irregular activity in the heart or require heart medication
  7. Have liver disease with symptoms
  8. Have history of hyponatremia (when you have decreased levels of sodium in the blood, which can cause confusion, seizures, fatigue and low levels of consciousness)
  9. Have history of hyperthermia (when you have a dangerously overheated body, usually in response to hot, humid weather)
  10. Weigh less than 48 kg
  11. Have recently engaged in suicidal behaviour or had serious suicidal thoughts (this will be assessed by the study team)
  12. Require ongoing therapy with a psychiatric medication
  13. Have a current eating disorder with active purging
  14. Have current major depressive disorder with psychotic features
  15. Are a serious risk to others
  16. Have recently received Electroconvulsive Therapy (ECT)
  17. Have recently engaged in ketamine-assisted therapy or used ketamine
  18. Have current substance use disorder with physiological dependence (not including caffeine or nicotine)
  19. Have recently used "Ecstasy" (material represented as containing MDMA)
  20. Are not able to give adequate informed consent
  21. Are not able to adhere to the requirements for procedures, attendance and timing of visits, and observe limits regarding study staff time and support as indicated by a time-limited clinical trial
  22. Are currently engaged in compensation litigation whereby financial gain would be achieved from prolonged symptoms of PTSD or any other psychiatric disorders
* Close Significant Other

  1. Meet criteria for PTSD
  2. Are pregnant or could become pregnant and not using birth control
  3. Have a history of, or a current psychotic disorder or bipolar 1 disorder or dissociative identity disorder
  4. Have a history of a medical condition that could make receiving MDMA unsafe (e.g. glaucoma, heart attack, stroke, aneurysm)
  5. Have a history of Diabetes Mellitus (Type 2) that a doctor determines is not stable
  6. Have hypothyroidism (low activity in the thyroid gland) and are not on thyroid replacement
  7. Have high blood pressure, a history of heart disease, heart failure, irregular activity in the heart or require heart medication
  8. Have liver disease with symptoms
  9. Have history of hyponatremia (when you have decreased levels of sodium in the blood, which can cause confusion, seizures, fatigue and low levels of consciousness)
  10. Have history of hyperthermia (when you have a dangerously overheated body, usually in response to hot, humid weather)
  11. Weigh less than 48 kg
  12. Have recently engaged in suicidal behaviour or had serious suicidal thoughts (this will be assessed by the study team)
  13. Require ongoing therapy with a psychiatric medication
  14. Have a current eating disorder with active purging
  15. Have current major depressive disorder with psychotic features
  16. Are a serious risk to others
  17. Have recently received Electroconvulsive Therapy (ECT)
  18. Have recently engaged in ketamine-assisted therapy or used ketamine
  19. Have current substance use disorder with physiological dependence (not including caffeine or nicotine)
  20. Have recently used "Ecstasy" (material represented as containing MDMA)
  21. Are not able to give adequate informed consent
  22. Are not able to adhere to the requirements for procedures, attendance and timing of visits, and observe limits regarding study staff time and support as indicated by a time-limited clinical trial
  23. Are currently engaged in compensation litigation whereby financial gain would be achieved from prolonged symptoms of PTSD or any other psychiatric disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure (FIM) | 3-Month Follow-up
  The Feasibility of Intervention Measure (FIM) is a self-report questionnaire in which respondents indicate the extent to which they believe that the treatment can be delivered in a given setting. Respondents indicate their responses on a five-point Likert-type (1=completely disagree, 5= completely agree).
Safety of Intervention | Baseline (enrolment) to Follow-up (3-month follow-up)
  Safety will be assessed by examining the frequency and severity of adverse events (AEs), serious AEs (SAEs), treatment emergent AES (TEAEs), and AEs of special interest. Participants are asked to report any AEs, SAEs, TEAEs, and AEs of special interest as they happen and during any communication with the therapist or independent assessor.
Intervention Appropriateness Measures (IAM) | 3-month follow-up
  Intervention Appropriateness Measures (IAM) is a self-report measure of the perceived fit, relevance, or compatibility of an intervention. Respondents record their answers on a five-point Likert-type scale (1=completely disagree, 5= completely agree).
Long Term Follow-Up Questionnaire (LTFUQ) | 3-Month Follow-up
  The Long Term Follow-Up Questionnaire (LTFUQ) is a self-report measure that assesses the long-term benefits and harms of MDMA-assisted therapy.
Clinician Administered PTSD Scale (CAPS-5) | Baseline (enrolment) to Follow-up (3-month follow-up)
  The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a clinician administered and scored assessment of PTSD symptoms via structured interview based upon PTSD diagnosis in DSM-5. It contains symptom subscales, a total severity score, and a diagnostic score. The total severity score is a sum of symptom frequency and intensity scores for the subscales B (re-experiencing), C (avoidance) and D (hypervigilance) and ranges from 0 to 136, with higher scores indicating greater severity of PTSD symptoms.

SECONDARY OUTCOMES:
Posttraumatic Stress Disorder Checklist for the DSM-5 (PCL-5) | Baseline (enrolment) to Follow-up (3-month follow-up)
  PTSD Checklist for the DSM-5 (PCL-5) is a self-report questionnaire in which respondents indicate the presence and severity of PTSD symptoms, derived from the DSM-5 symptoms of PTSD. Participants indicate how much distress they have experienced due to symptoms on a five-point Likert-type scale (1 = not at all, 5 = extremely). The total PCL-5 score (a sum of all 20 items) provides an index of overall PTSD symptom severity with higher scores indicating higher severity.
Quality of Relationships Inventory (QRI) | Baseline (enrolment) to Follow-up (3-month follow-up)
  The Quality of Relationships Inventory (QRI) is a self-report questionnaire that uses the role of situational, intrapersonal, and interpersonal in social support processes to assess supportive and conflictual aspects of close non-intimate relationships.
Couple Satisfaction Index (CSI) | Baseline (enrolment) to Follow-up (3-month follow-up)
  The Couple Satisfaction Index (CSI) is a self-report questionnaire that measures intimate relationship functioning. Respondents answer most of the questions on a six-point Likert-type scale (0= never, 5= all the time) and one question on a seven-point Likert-type scale ( 0= extremely unhappy, 6= perfect).
Patient Health Questionnaire-9 (PHQ-9) | Baseline (enrolment) to Follow-up (3-month follow-up)
  The Patient Health Questionnaire-9 (PHQ-9) is used to assess depressive symptom severity. The PHQ-9 includes items which correspond with the diagnostic criteria for DSM-IV major depressive disorder. Scores can indicate either no depression, minimal, mild, moderate, moderately severe, or severe depression. Higher scores indicate higher severity in depressive symptoms.

OTHER OUTCOMES:
Posttraumatic Growth Inventory (PTGI) | Baseline (enrolment) to Follow-up (3 month follow-up)
  The Posttraumatic Growth Inventory (PTGI) is a 21-item self-report measure of perceived growth or benefits occurring after a traumatic event. It contains five subscales: relationship to others, new possibilities, personal strength, spiritual change, and appreciation of life.
Self-Compassion Scale-Short Form (SCS-SF) | Baseline (enrolment) to Follow-up (3-month follow-up)
  The Self-Compassion Scale-Short Form (SCS-SF) is a 12-item self-report measures that assess self-compassion. This measure is comprised of the following subscales: self-kindness, self-judgement, common humanity, isolation, mindfulness, and over-identification. Respondents answer questions on a five-point Likert-type scale (1= almost never, 5= almost always).
Brief Experiential Avoidance Questionnaire (BEAQ) | Baseline (enrolment) to Follow-up (3-month follow-up)
  The Brief Experiential Avoidance Questionnaire (BEAQ) is a 15-item self-report measure that assesses experiential avoidance. Respondents rate the extent to which they agree with each item on a six-point Likert-type scale (1 = strongly disagree, 6= strongly agree).
Alcohol Use Disorders Identification Test (AUDIT), Cannabis Use Disorders Identification Test-Revised (CUDIT-R), and Drug Use Disorders Identification Test (DUDIT) | Baseline (enrolment) to Follow-up (3-month follow-up)
  The Alcohol Use Disorders Identification Test (AUDIT), Cannabis Use Disorders Identification Test-Revised (CUDIT-R), and Drug Use Disorders Identification Test (DUDIT) are self-report questionnaires that assess alcohol and substance use.
Brief Posttraumatic Cognitions Inventory (PTCI-9) | Baseline (enrolment) to Follow-up (3-month follow-up)
  The Brief Posttraumatic Cognitions Inventory (PTCI-9) is a nine-item self-report questionnaire that measures appraisals related to trauma. Respondents answer the questionnaire on a seven-point Likert-type scale (1= totally disagree, 7= totally agree).
MOS Social Support Survey (MOS-SSS) | Baseline (enrolment) to Follow-up (3-month follow-up)
  The MOS Social Support Survey (MOS-SSS) is a 20-item multidimensional self-report questionnaire that assess perceived availability of social support. Respondents answer questions on a seven-point Likert-type scale (1 = none of the time, 7= all of the time), where higher score indicate greater levels of available social support.
Significant Others' Responses to Trauma Scale (SORTS) | Baseline (enrolment) to Follow-up (3-month follow-up)
  The Significant Others' Responses to Trauma Scale (SORTS) is a 14-item self-report questionnaire that measures relationship problems and the psychological distress of partners of people with PTSD. Respondents answer questions on a five-point Likert scale (0-4).
Modified Experiences in Close Relationships (ECR-M16) | Baseline (enrolment) to Follow-up (3-month follow-up)
  The Modified Experiences in Close Relationships (ECR-M16) is a 16-item self-report questionnaire that assesses attachment style. Half of the items on the scale measure attachment anxiety and the other half measures attachment avoidance. Respondents answer questions on a seven-point Likert-type scale (1= disagree, 7=agree).
Psychological Insights Questionnaire (PIQ) | Baseline (enrolment) to Follow-up (3-month follow-up)
  The Psychological Insights Questionnaire (PIQ) is a a 23-item self-report measure that assesses acute experiences of insight (i.e., beliefs, memories, emotions, etc.). Respondents answer questions on a six-point Likert-type scale (0= no, not at all; 5= extremely).
Mystical Experiences Questionnaire (MEQ30) | Baseline (enrolment) to Follow-up (3-month follow-up)
  The Mystical Experiences Questionnaire (MEQ30) is a 30-item self-report questionnaire that assesses discrete mystical experiences. Respondents rate the extent to which the experience mystical feeling, positive mood, transcendence of space/time, and ineffability on a five-point Likert-type scale (0= no/not at all, 4= extreme).
Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline (enrolment) to Follow-up (3-month follow-up)
  The Columbia-Suicide Severity Rating Scale (C-SSRS) is a clinician-administered measure of suicidal behaviour devised to detect potential suicidal thoughts or behaviours. It is designed to assess suicidal ideation, ideation intensity, and behaviour.
Credibility Expectancy Questionnaire (CEQ) | Baseline (enrolment)
  The Credibility Expectancy Questionnaire (CEQ) is a six-item self-report measure of beliefs about treatment credibility and expectancy of treatment outcomes. The some questions on the questionnaire are answered on a scale ranging from 1 (not at all) to 9 (very much) and that others are answered on a scale ranging from 0 (not at all) to 100% (very much).
Working Alliance Inventory-Observer Form (WAI-O) | First therapy session, Mid-point, and Follow-up (3-month follow-up)
  The Working Alliance Inventory-Observer Form (WAI-O) is a 36-item observer-rated measure of the alliance between a therapist and client. Observers rate each item on a scale from 1 (Never applies to the dyad) to 7 (Always applies to the dyad).

CONTACTS AND LOCATIONS:
Overall Officials: Paul Uy, MD, Principal Investigator — Remedy Institute; Anne Wagner, PhD, Study Chair — Remedy Institute
Locations (1):
- Remedy Institute, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No